CLINICAL TRIAL: NCT01096758
Title: 5-year Follow-up of the Comparison of Life and Physical Health in Adult Patients With PKU and Healthy Age Matched Controls
Brief Title: Follow-up of Adult Phenylketonuria (PKU) Patients
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Koletzko - Office, Prof., Ludwig-Maximilians - University of Munich
Other Study IDs: A-PKU2010
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Nutritional Deficiencies; Phenylketonuria
Keywords: PKU; phenylketonuria; adult; patient; development; nutritional deficiencies; neurological outcome; psychological and neurological development; comparison with healthy adults; longitudinal development; quality of life
MeSH Terms: conditions — Malnutrition; Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood cheek cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PKU patients
- healthy controls

SUMMARY:
Adult patients with phenylketonuria (PKU) at the age around 40 years belong to the first patients generation with early treatment of the disease. PKU is caused by an inborn error of the amino acid metabolism and the so far best suitable therapy is an early and strict diet, which is low in phenylalanine.

Besides an early and continuously treatment in childhood, the nutritional and medical support during adolescence and adulthood have been suggested to influence the long-term physical health of adult PKU patients. As many adult PKU patients tend to neglect the necessarily strict diet, they do not get a balanced diet. For PKU patients some nutrients, which may be rare in an unbalanced diet, might help to improve health status, physical and neurological performance and quality of life.

Information about the longitudinal development of the patients status and the influence of the type of their medical care is not available. In this 5 year follow-up the investigators aim to study the quality of life and the medical, nutritional and psychological status of adult PKU patients, in whom corresponding information has already been collected previously.

ELIGIBILITY:
Inclusion Criteria:

* assured clinical diagnose of PKU or proof of mutation in the phenylalanine hydroxylase gene (for PKU patients only)
* both groups need to hand in a signed consent to participate in the study
* controls: have to be omnivores and should not be on drugs, which influence the lipid metabolism, during the last 3 months
* attendance of the last study trial

Exclusion Criteria:

* not fulfill the inclusion criteria

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult PKU patients who are or have been attending the Departements of Metabolic Diseases of the Klinikum der Universität München will be recruited for this study, if they had been participating already in the last study trial comparing adult PKU patients with healthy controls.
  It will be attempted to include the same control persons as in the last study trial.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Dr. von Hauner Childrens Hospital, München, Germany